CLINICAL TRIAL: NCT02136147
Title: Naturalistic Study of ADHD Medication and Predictors of Treatment Outcome
Brief Title: ADHD Medication and Predictors of Treatment Outcome
Acronym: ADAPT
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Linda Halldner Henriksson, MD, PhD, Karolinska Institutet
Other Study IDs: ADAPT; LS 1110-1339 (Other Grant/Funding Number: ALF/PPG); SLS-309701 (Other Grant/Funding Number: Stiftelsen Söderström-Königska sjukhemmet)
Record Dates: First submitted 2014-04-30; First posted 2014-05-12 (Estimated); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Attention Deficit Disorder With Hyperactivity (ADHD)
Keywords: Attention Deficit Disorder with Hyperactivity; Neuropsychiatry; Drug therapy; Pharmacogenetics; Child Psychiatry
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; Atomoxetine Hydrochloride; Lisdexamfetamine Dimesylate; Guanfacine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Children with ADHD medication: Identified responders and non-responders in children/adolescents starting medication for treatment of ADHD in public child and adolescent psychiatric services in Stockholm, on Gotland, and in Västerbotten.
  Interventions: Drug: methylphenidate medication; Drug: atomoxetine medication; Drug: lisdexamphetamine medication; Drug: guanfacine medication
- Lisdexamphetamine medication: Identified responders and non-responders in children/adolescents starting medication with lisdexamphetamine in public child and adolescent psychiatric services in Stockholm and on Gotland.
  Interventions: Drug: lisdexamphetamine medication
- Atomoxetine medication: Identified responders and non-responders in children/adolescents starting medication with atomoxetine in public child and adolescent psychiatric services in Stockholm and on Gotland.
  Interventions: Drug: atomoxetine medication
- Methylphenidate medication: Identified responders and non-responders in children/adolescents starting medication with methylphenidate in public child and adolescent psychiatric services in Stockholm and on Gotland.
  Interventions: Drug: methylphenidate medication
- Guanfacine medication: Identified responders and non-responders in children/adolescents starting medication with guanfacine in public child and adolescent psychiatric services in Stockholm and on Gotland.
  Interventions: Drug: guanfacine medication

INTERVENTIONS:
Drug: methylphenidate medication
  Other Names: N06BA04; Concerta; Ritalin; Equasym; Medikinet
  Groups: Children with ADHD medication; Methylphenidate medication
Drug: atomoxetine medication
  Other Names: N06BA09; Strattera
  Groups: Atomoxetine medication; Children with ADHD medication
Drug: lisdexamphetamine medication
  Other Names: N06BA12; Elvanse
  Groups: Children with ADHD medication; Lisdexamphetamine medication
Drug: guanfacine medication
  Other Names: C02AC02; Intuniv
  Groups: Children with ADHD medication; Guanfacine medication

SUMMARY:
ADHD medication of children and adolescents is becoming increasingly common. Clinical experience and scientific studies have proven that approximately 30% of children/adolescents with ADHD do not benefit from this treatment. However, there is insufficient knowledge about who these children are. All children and adolescents, who start treatment with ADHD medication at public Child and Adolescent Psychiatry units in Stockholm, on Gotland, an in Västerbotten, will be asked to participate in the study. The investigators intend to monitor the patients´clinical symptoms and possible side-effects after treatment start. The investigators will collect background information and saliva samples from the patient and his/her parents to be able to study if there are any genetic (hereditary) or other markers that can predict positive or negative outcomes of the ADHD medication. With this information, the investigators aim at, to a greater extent, be able to individualize treatment choices for children and adolescents with ADHD without unnecessary, costly and possibly unfavorable treatment attempts.

DETAILED DESCRIPTION:
The specific aims for the ADAPT study are:

1. Investigate if certain gene polymorphisms are associated with poor effect of ADHD drugs (non-responders).
2. Investigate if other biologically, phenotypic or psychosocial factors are associated with poor effect of ADHD drugs (non-responders).
3. Investigate if the frequency of side-effects of ADHD drugs differs between children with different genotypes.
4. Investigate if the frequency of side-effects of ADHD drugs differs between children with different phenotypic and/or psychosocial factors

Method:

This study has a naturalistic design. The aim is to map all new treatments with ADHD drugs at all 13 public BUP units in Stockholm County, one BUP unit on Gotland, and three BUP units in Västerbotten Region. The participation means that medication is initiated as planned in normal clinical practice by the child´s ordinary physician, and beyond this only means a somewhat denser and more structured follow-up. In addition, the investigators will ask for saliva samples from the patient and his/her parents. The investigators aim at including at least 1000 individuals in total in the study.

Part of the data will be collected via the national Quality Register for ADHD Treatment Follow-up (BUSA), which has approved security procedures approved by the Swedish Data Inspection Board.

Case report forms are computerized and separate from the database registry for collected study data. The database and detailed variable lists are constructed in collaboration with professional database managers.

Standard Operation Procedures are designed in collaboration by project coordinator, study nurse and principal investigator, and may be revised after pilot phase.

Collected samples will be stored at KI biobank.

Data analysis:

1. To judge if the patient is a responder to ADHD drugs the SNAP-IV rating of ADHD symptoms (before and after medication start) is used. The patients who at 3 months have an at least 40% reduction in SNAP-IV score are reckoned "responders" and those who at the same time point have a less than 20% change in SNAP-IV score are reckoned "non-responders". Differences between the groups will be analyzed with logistic regression, with responder status as depending variable, and genotype and the other risk markers (biological, phenotypic, and psychosocial markers) as independent variables after correction for symptoms at baseline. Even a 50% drop-out rate will (i.e. 1000 out of estimated 2000 eligible individuals) give a 98% power to identify a 49% increase in non-responder proportion for a specific genotype.
2. Concomitantly, the outcome in side-effects, heart rate, blood pressure, weight (z-score) and length (z-score) will be analyzed with linear regression with the same independent variables.
3. The analyses are performed separately for each ADHD drug.
4. There are significantly more boys than girls (about 4:1) with ADHD. Given the sex difference in prevalence it is obvious to also include sex as a covariate in our analyses of treatment outcome.
5. Missing data will be treated according to the principles of complete case and multiple imputation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ADHD
* Starting medication against ADHD symptoms with atomoxetine, methylphenidate, lisdexamphetamine, or guanfacine

Exclusion Criteria: Any medication against ADHD the last 3 months

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children/adolescents starting ADHD medication at the public child and adolescent psychiatry services in Stockholm and on Gotland
Sampling Method: Non-Probability Sample
Enrollment: 632 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2021-07 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
change in SNAP-IV Teacher and Parent rating scale (Swanson, Nolan and Pelham ADHD Rating Scale) | at 3 months follow-up
  ADHD symptoms
change in P-SEC (Pediatric Side Effects Checklist) | at 3 months follow-up
  Side-effect measure

SECONDARY OUTCOMES:
change in C-GAS (Children´s global assessment scale) | at 12 months follow-up
  global functioning measure
change in CGI-S (Clinical Global Impression- of Severity) | at 12 months follow-up
  disease severity
change in SNAP-IV Teacher and Parent rating scale | at 1 month follow-up
  ADHD symptoms
change in SNAP-IV Teacher and Parent rating scale | at 6 months follow-up
  ADHD symptoms
change in SNAP-IV Teacher and Parent rating scale | at 12 months follow-up
  ADHD symptoms
change in P-SEC (Pediatric Side Effects Checklist) | at 1 month follow-up
  side effect measure
change in P-SEC (Pediatric Side Effects Checklist) | at 6 months follow-up
  side effect measure
change in P-SEC (Pediatric Side Effects Checklist) | at 12 months follow-up
  side effect measure
change in Spence Children's Anxiety Scale (SCAS) | at 1 month follow-up
  symptoms of anxiety
change in Spence Children's Anxiety Scale (SCAS) | at 3 months follow-up
  symptoms of anxiety
change in Spence Children's Anxiety Scale (SCAS) | at 6 months follow-up
  symptoms of anxiety
change in Spence Children's Anxiety Scale (SCAS) | at 12 months follow-up
  symptoms of anxiety
change in heart rate | at 1 month follow-up
change in heart rate | at 3 months follow-up
change in heart rate | at 6 months follow-up
change in heart rate | at 12 months follow-up
change in systolic blood pressure | at 1 month follow-up
change in systolic blood pressure | at 3 months follow-up
change in systolic blood pressure | at 6 months follow-up
change in systolic blood pressure | at 12 months follow-up
change in diastolic blood pressure | at 1 month follow-up
change in diastolic blood pressure | at 3 months follow-up
change in diastolic blood pressure | at 6 months follow-up
change in diastolic blood pressure | at 12 months follow-up
change in weight z-score | at 1 month follow-up
change in weight z-score | at 3 months follow-up
change in weight z-score | at 6 months follow-up
change in weight z-score | at 12 months follow-up
change in height z-score | at 6 months follow-up
change in height z-score | at 12 months follow-up
change in Autism Spectrum Screening Questionnaire (ASSQ) score | at 3 months follow-up
  symptoms of autism
change in Autism Spectrum Screening Questionnaire (ASSQ) score | at 1 months follow-up
  symptoms of autism
change in Autism Spectrum Screening Questionnaire (ASSQ) score | at 6 months follow-up
  symptoms of autism
change in Autism Spectrum Screening Questionnaire (ASSQ) score | at 12 months follow-up
  symptoms of autism

OTHER OUTCOMES:
change in self-harm frequency | at 12 months follow-up
  change in self-harm frequency behavior as noted in the quality register BUSA
change in suicide attempt frequency | at 12 months follow-up
  change in suicide attempt frequency as reported in quality register BUSA

CONTACTS AND LOCATIONS:
Locations (1):
- Division for Child and Adolescent Psychiatry in Stockholm, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lilja MM, Lichtenstein P, Serlachius E, Bhagia J, Malmberg K, Malm C, Lenhard F, Halldner L. Can response to ADHD medication be predicted? Eur Child Adolesc Psychiatry. 2025 Aug;34(8):2431-2442. doi: 10.1007/s00787-025-02650-8. Epub 2025 Jan 29. PMID 39875602
- [Derived] Lilja MM, Sandblom E, Lichtenstein P, Serlachius E, Hellner C, Bhagia J, Halldner L. The effect of autistic traits on response to and side-effects of pharmacological ADHD treatment in children with ADHD: results from a prospective clinical cohort. J Neurodev Disord. 2022 Mar 6;14(1):17. doi: 10.1186/s11689-022-09424-2. PMID 35249540